CLINICAL TRIAL: NCT00571337
Title: Prospective Study of Predictive Factors of Sustained Remission of Crohn's Disease After Stopping Infliximab
Brief Title: Stop Infliximab in Patients With Crohn's Disease
Acronym: STORI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Responsible Party: LEMANN MARC, getaid
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GETAID 2005-1
Record Dates: First submitted 2007-07-25; First posted 2007-12-12 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-07

CONDITIONS: Crohn Disease
Keywords: Stop infliximab.
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Infliximab — Stopping infliximab in patients having been treated with this drug for at least one year and in stable remission for at least 6 month.

SUMMARY:
1 Project summary 1.1 Rational. Accent 1 study has demonstrated the superiority of Infliximab over placebo in a systematic treatment strategy of Crohn 's disease every 8 weeks during one year. However the optimal strategy beyond one year of treatment is not established. Particularly, the need for carrying on systematic treatment with infliximab in all the patients has not been demonstrated.

1.2 Primary objective. Determine factors associated with a low risk of clinical relapse after stopping infliximab in CD patients in remission (CDAI<150) and regularly treated with infliximab for at least one year.

1.3 Main objective and main judgement criteria. Determine predictive factors for relapse within one year after stopping infliximab. Main judgement criteria is the clinical relapse after stopping infliximab. Clinical relapse is defined either by a CDAI>250 or by a CDAI between 150 and 250 if this CDAI is confirmed over two consecutive weeks with an increase of at least 70 points over baseline for the two consecutive measures.

1.4 Secondary objectives and judgement criteria. Determine the time to-relapse Determine predictive factors for short-term relapse (<2 months)after stopping infliximab.

Determine response to infliximab retreatment in these patients. Determine tolerance to infliximab retreatment in these patients. Determine predictive factors for an absence of response to retreatment. Determine predictive factors for infliximab retreatment intolerance. Determine sustained response in the retreated patients.

1.5 Type of study Open-label prospective study of stopping regular treatment. Inclusion period: minimum one year, possibly prolonged to reach 100 patients. Patients will be followed up every two months for at least 18 months after stopping infliximab.

1.6 Justification of the number of patients Number of patients to include is at least 100. This recruitment should be reached within one year. This number should allow to disclose predictive factors associated with a relative risk of at least 2 if this factor is equilibrated (50% at risk patients) or 3 is this factor is disequilibrated (90% at risk patients).

ELIGIBILITY:
Inclusion criteria:

* Crohn's disease.
* Age > 18 years.
* Patient written informed consent.
* Patient having been treated with infliximab for confirmed Crohn's disease with active intestinal lesions.
* Patient treated with infliximab for at least 1 year, associated with an immunosuppressor for at least one year, with a maximum interval between 2 infliximab infusions of 3 months.
* Patient with continuous remission without steroids for at least 6 months, except IV steroids for infusion reaction prophylaxis.
* CDAI<150.
* Contraception all over the study.

Exclusion criteria:

* Patient having experienced an severe acute infusion reaction to infliximab, defined by an anaphylactoïd reaction (drop in blood pressure, bronchospasm, dyspnea) requiring the arrest of the infliximab infusion.
* Patient having experienced a severe delayed infusion reaction to infliximab, defined by fever, arthralgia, myalgia, requiring a steroid treatment.
* Patient with dominant perianal disease and absence of active intestinal disease at the time of infliximab induction.
* Patient with active perianal disease at the time of inclusion.
* Patient with stoma.
* Patient with debilitating extra-intestinal manifestation at the time of inclusion.
* Non cooperating subjects.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2005-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Relapse of Crohn's disease assessed by a CDAI > 250 or a CDAI between 150 and 250 at two consecutive weeks, with an increase of at least 70 points over baseline. | Time to relapse over one year
Evaluation of demographic, clinical and endoscopic factors predictive of relapse of Crohn's disease after stopping infliximab, with univariate and multivariate analysis. | Factors influencing time to relapse over one year.

SECONDARY OUTCOMES:
Tolerance and safety of infliximab retreatment in patients experiencing a relapse. | Follow up over 4 months including 3 infliximab retreatment s.
predictive factors of short term-relapse (<2 months) after stopping infliximab, in the follow up of the patients. | at least 12 month and a maximum of 18 months.
Clinical response to infliximab retreatment, assessed 4 weeks after retreatment using CDAI. A clinical response is defined by a 70 points drop (and at least 25%) as compared to relapse CDAI. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Louis Edouard, PhD, Principal Investigator — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives
Locations (23):
- Belgium (2):
  - Gent University Hospital, Ghent
  - CHU LIEGE - Sart Tilman, Liège
- France (21):
  - Chu Amiens, Amiens
  - Chu Besancon, Besançon
  - Hopital Saint Andre, Bordeaux
  - CHU CAEN, Caen
  - Hopital Beaujon, Clichy
  - Hopital Louis Mourier, Colombes
  - Hopital Henri Mondor, Créteil
  - CHRU Lille, Lille
  - Chu Marseille - Hopital Nord, Marseille
  - Ch Le Raincy Montfermeil, Montfermeil
  - Chu Montpellier, Montpellier
  - Chu Nantes, Nantes
  - Hopital Lariboisiere, Paris
  - Hopital Saint Louis, Paris
  - Hopital Georges Pompidou, Paris
  - Hopital Haut Leveque, Pessac
  - CHU LYON, Pierre-Bénite
  - Chu Rouen, Rouen
  - Chu Strasbourg, Strasbourg
  - Chu Toulouse, Toulouse
  - Chu Tours, Tours

REFERENCES:
- [Background] Vermeire S, Louis E, Carbonez A, Van Assche G, Noman M, Belaiche J, De Vos M, Van Gossum A, Pescatore P, Fiasse R, Pelckmans P, Reynaert H, D'Haens G, Rutgeerts P; Belgian Group of Infliximab Expanded Access Program in Crohn's Disease. Demographic and clinical parameters influencing the short-term outcome of anti-tumor necrosis factor (infliximab) treatment in Crohn's disease. Am J Gastroenterol. 2002 Sep;97(9):2357-63. doi: 10.1111/j.1572-0241.2002.05991.x. PMID 12358256
- [Background] Parsi MA, Achkar JP, Richardson S, Katz J, Hammel JP, Lashner BA, Brzezinski A. Predictors of response to infliximab in patients with Crohn's disease. Gastroenterology. 2002 Sep;123(3):707-13. doi: 10.1053/gast.2002.35390. PMID 12198696
- [Background] Farrell RJ, Alsahli M, Jeen YT, Falchuk KR, Peppercorn MA, Michetti P. Intravenous hydrocortisone premedication reduces antibodies to infliximab in Crohn's disease: a randomized controlled trial. Gastroenterology. 2003 Apr;124(4):917-24. doi: 10.1053/gast.2003.50145. PMID 12671888
- [Background] Baert F, Noman M, Vermeire S, Van Assche G, D' Haens G, Carbonez A, Rutgeerts P. Influence of immunogenicity on the long-term efficacy of infliximab in Crohn's disease. N Engl J Med. 2003 Feb 13;348(7):601-8. doi: 10.1056/NEJMoa020888. PMID 12584368
- [Background] Tampo Y, Yonaha M. Antioxidant mechanism of Mn(II) in phospholipid peroxidation. Free Radic Biol Med. 1992;13(2):115-20. doi: 10.1016/0891-5849(92)90072-o. PMID 1516837
- [Background] Parsi MA, Lashner BA. Safety of infliximab: primum non nocere. The safety profile of infliximab in patients with Crohn's disease: the Mayo Clinic experience in 500 patients. Inflamm Bowel Dis. 2004 Jul;10(4):486-7. doi: 10.1097/00054725-200407000-00028. No abstract available. PMID 15475765
- [Background] Keane J, Gershon S, Wise RP, Mirabile-Levens E, Kasznica J, Schwieterman WD, Siegel JN, Braun MM. Tuberculosis associated with infliximab, a tumor necrosis factor alpha-neutralizing agent. N Engl J Med. 2001 Oct 11;345(15):1098-104. doi: 10.1056/NEJMoa011110. PMID 11596589
- [Derived] Pierre N, Huynh-Thu VA, Baiwir D, Mazzucchelli G, Fleron M, Trzpiot L, Eppe G, De Pauw E, Laharie D, Satsangi J, Bossuyt P, Vuitton L, Vieujean S, Colombel JF, Meuwis MA, Louis E; GETAID and the SPARE-Biocycle research group. External validation of serum biomarkers predicting short-term and mid/long-term relapse in patients with Crohn's disease stopping infliximab. Gut. 2024 Nov 11;73(12):1965-1973. doi: 10.1136/gutjnl-2024-332648. PMID 39134391
- [Derived] Louis E, Mary JY, Vernier-Massouille G, Grimaud JC, Bouhnik Y, Laharie D, Dupas JL, Pillant H, Picon L, Veyrac M, Flamant M, Savoye G, Jian R, Devos M, Porcher R, Paintaud G, Piver E, Colombel JF, Lemann M; Groupe D'etudes Therapeutiques Des Affections Inflammatoires Digestives. Maintenance of remission among patients with Crohn's disease on antimetabolite therapy after infliximab therapy is stopped. Gastroenterology. 2012 Jan;142(1):63-70.e5; quiz e31. doi: 10.1053/j.gastro.2011.09.034. Epub 2011 Sep 22. PMID 21945953